CLINICAL TRIAL: NCT05307185
Title: A Comparison Among the Effects of the Low FODMAP Diet, a Tritordeum Based Diet, and Dietary Advice on the Gastrointestinal Symptom Profile in Patients With Irritable Bowel Syndrome-Diarrhea Variant (IBS-D): a Randomized Controlled Trial
Brief Title: Tritordeum-based Foods for IBS Symptoms
Acronym: TritoinIBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Francesco Russo, Coordinating Medical Director Functional GI Disorders Research Group, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRITOIBS22
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Diarrhea; Diet; FODMAPs; Tritordeum; Intestinal permeability; Symptoms; Dysbiosis; Gluten
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea; Dysbiosis

STUDY DESIGN:
Intervention Model Description: Multi-disciplinary, single-blind, parallel-group randomized controlled trial design
Who Masked: Participant
Masking Description: The investigator, but not the patients will know the real identity of the treatment assignment (food preparation and packaging will be unlabelled and not recognizable).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tritordeum-based Food (TBD) (Experimental): A controlled TBD will be provided to each patient. The daily menu will be breakfast, mid-morning snacks, lunch, afternoon snacks, and dinner. This intervention diet implies that each patient in the study has to consume flour, bread, breakfast biscuits, taralli, and pasta prepared exclusively with Tritordeum. The diets will be designed by matching basal metabolism and daily energy consumption with anthropometric data of all patients to assign suitable and tailored dietary regimens. The software utilized to assess the daily intake of macronutrients (50% carbohydrates, 30% lipids, and 20% proteins) will be the same as LFD.
  Interventions: Dietary Supplement: Tritordeum-based food
- Low-FODMAPs diet (LFD) (Active Comparator): A personalized LFD will be assigned after reviewing a food diary and having a one-on-one personal consultation with a nutritionist. Diet will match the basal metabolic rate and daily energy expenditure. A detailed weekly structured menu based on three meals (breakfast, lunch, and dinner) and two snacks (morning and afternoon) will be provided. Patients also will receive a booklet detailing what foods are allowed, which foods to avoid and which foods to reduce based on the classifications used by Monash University and cut-off values for each FODMAPs subgroup. Nutritionists have already created a leaflet for patients in the study with details on where to buy specific products. Besides, nutritionists will guarantee adequate fiber intake, also offering advice on cooking without onions and garlic and other high-FODMAP foods. Drinking alcohol will not be recommended, although it is not high in FODMAPs.
  Interventions: Dietary Supplement: Tritordeum-based food
- Specific dietary advice for IBS (Active Comparator): According to NICE BDA Irritable bowel syndrome dietary advice, a controlled diet will be provided. All the food items (bread, pasta, "taralli" - local salty biscuits, and breakfast biscuits) will be prepared using durum wheat flour commercially available and anonymized to guarantee masking. Dietary recommendations include eating slowly, limiting alcohol, spicy food and fatty foods, caffeine, carbonated drinks; avoiding chewing gums and sweeteners containing polyols; small and frequent meals, stressful conditions.
  Interventions: Dietary Supplement: Tritordeum-based food

INTERVENTIONS:
Dietary Supplement: Tritordeum-based food — Diets will last 12 weeks with intermediate nutritional checks every four weeks before returning to the final study visit.

SUMMARY:
People with irritable bowel syndrome (IBS), especially those with diarrhea (IBS-D), often describe worsening symptoms after eating certain foods. A structured dietary approach may represent a reliable strategy to improve their symptoms. In this framework, the diet low in oligosaccharides, disaccharides, monosaccharides, and fermentable polyols (FODMAPs - LFD) has been demonstrated to mitigate symptoms and reduce inflammatory status, increase vitamin D content, and affect the lipidomic profile. Unfortunately, adherence to LFD can be somewhat problematic, needing continuous nutritional support. Other dietary approaches with putative beneficial effects have been proposed to overcome these limitations. Among them, Tritordeum-based foods (TBD, bread, bakery products, and pasta) in substitution of other cereals seem to achieve promising results. TBD may represent a valid alternative, with high palatability, especially among Italian patients for whom pasta is considered one of the main assets of dietetic culture and easier to manage in their daily habits. Given these premises, this study aims to evaluate, in a randomized single-blinded controlled trial, the effects of 12-weeks of TBD compared with LFD and dietary advice of the same duration in improving the symptom profile well as the intestinal permeability and reducing putative dysbiosis of IBS-D patients. Along with the clinical study, an evaluation of gluten and proteomic composition will be performed to examine more in detail the intrinsic characteristics of Tritordeum.

DETAILED DESCRIPTION:
A structured dietary approach could represent a reliable alternative strategy to treat patients with functional gastrointestinal disorders such as irritable bowel syndrome (IBS), mainly in its diarrhea variant (IBS-D). It is now well established that many people with IBS often describe worsening symptoms eating certain foods, such as those containing fermentable oligosaccharides, disaccharides, monosaccharides, and polyols (FODMAPs). These short-chain carbohydrates are present in some foods, including wheat and beans. They may contribute to different digestive symptoms such as bloating, abdominal pain, and diarrhea due to poor absorption in the small intestine. In this way, FODMAPs are digested by colonic bacteria, releasing gas in the colon.

Furthermore, FODMAPs can act as osmotic agents, increasing the water volume in the stool. In the last years, our group has focused research on the properties of a low FODMAPs diet (LFD) in the clinical management of patients with IBS-D, demonstrating that these patients benefit from a 12 weeks-LFD in mitigating the symptoms, reducing the inflammatory status, increasing the vitamin D content, and affecting the lipidomic profile. Unfortunately, adherence to LFD can be somewhat problematic, needing continuous nutritional support.

Actually, alternative dietary approaches for these disorders may be hypothesized. It is now well established that, beyond non-celiac wheat sensitivity (NCWS), many individuals suffering from IBS-D or generical gluten-related disorders and mainly complainIng of abdominal bloating seem to benefit from removing wheat from the diet.

The multifaceted setting of nutrients in wheat-based foods, other than gluten, could account for the different IBS symptoms. It has already been postulated that some monococcal diploid grain lines, with minimal activation of the innate immunity and a reduced amount of toxic gluten peptides, could be helpful for IBS-D patients. Among them, alternative grains such as Tritordeum seem to achieve good results. Tritordeum is a cereal derived from durum wheat and wild barley hybridization. Originally cultivated with traditional techniques in Spain, it has more recently grown in Apulia, a southern Italy region. Tritordeum grows well with little care, even in adverse conditions. Noteworthy, this cereal has significantly lower levels of gliadins, fewer carbohydrates and fructans, and a higher content of dietary fibers, proteins, and antioxidants than classic wheat. However, the presence of gluten makes this cereal not suitable for celiac patients.

Thus, cereals such as Tritordeum, once further characterized in their proteomic profile and gluten composition, could offer opportunities for an innovative nutritional approach for patients suffering from IBS and, more in general, wheat-related disorders. Our group recently performed a pilot study to investigate the effects of a 12-week diet with Tritordeum-based foods (bread, bakery products, and pasta) in substitution of other cereals on the GI symptoms and the status of the GI barrier in IBS-D patients. This diet proved to reduce the patients' symptoms by affecting intestinal permeability significantly. The purpose of this study is to evaluate, in a randomized controlled trial, the beneficial effects of 12-weeks of TBD compared with LFD or specific advice for IBS of the same duration in improving the symptom profile of IBS-D patients.

ELIGIBILITY:
Inclusion Criteria:

* Rome IV criteria for IBS diarrhea variant (IBS-D).
* Low-lactose diet is allowed, provided that patients agree to keep this intake constant throughout the study period, except in the case of randomization in the treatment arm with a low-FODMAPs diet.
* The use of probiotic products is permitted, and patients who consume probiotic products must be instructed to continue taking the same amount previously taken throughout the study period.
* The drugs used to treat IBS, including antidepressants, will be admitted provided they are used regularly and have a stable dosage for at least one month prior to inclusion in the study.
* Patients must be willing to change their current diet to participate in the study for the whole study period.

Exclusion Criteria:

* Serious cardiac, hepatic, neurological or psychiatric diseases.
* GI diseases other than IBS (e.g., inflammatory bowel disease, celiac disease) that could explain current symptoms.
* Patients who previously had a low-content diet of particular substances (for example, low FODMAPs content, vegan diet, a gluten-free diet). - This last category of subjects will be able to return to the study provided they suspend the gluten-free diet until the symptoms reappear.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in the total score of the irritable bowel syndrome - severity scoring system (IBS-SSS) questionnaire | Before the start of the study (time 0) and after 90 days of treatment (time 90).
  IBS-SSS contains 5 specific questions with instructions on how to score them. Each of the five questions (pain severity, pain frequency, abdominal distension severity, bowel movement satisfaction, quality of life) ranges from 0 to a maximum score of 100 using a visual analog scale (VAS), leading to a total possible score of 500.
  The primary outcome corresponds to a change in the total score of the IBS-SSS questionnaire at the end of the treatment period compared to baseline, and the proportion of patients who will achieve a difference in the total symptom score of IBS-SSS ≥50 after diet. Such difference is considered a significant clinical improvement.

SECONDARY OUTCOMES:
Change in the score of the single symptom items of the irritable bowel syndrome - severity scoring system (IBS-SSS) questionnaire | Before the start of the study (time 0) and after 90 days of treatment (time 90).
  IBS-SSS contains 5 specific questions with instructions on how to score them. Each of the five questions (pain severity, pain frequency, abdominal distension severity, bowel movement satisfaction, quality of life) ranges from 0 to a maximum score of 100 using a visual analog scale (VAS). The secondary outcome is the measure of the effects of the dietary interventions on the individual symptom items score of IBS-SSS, as well as on the characteristics of the stool habit through the administration of the diaries.
Change in the psychological symptom profile evaluated by Symptom Checklist-90- Revised (SCL-90-R) | Before the start of the study (time 0) and after 90 days of treatment (time 90).
  The Symptom Checklist-90- Revised (SCL-90-R) questionnaire is one of the best-known and most used self-report measures in the psychopathological field. SCL-90-R evaluates a broad spectrum of psychopathological symptoms, namely nine primary symptom dimensions and three global indices. Only the Global Severity Index (GSI), the best indicator of the current intensity of psychic distress perceived by the subject will be considered. The raw scores will be transformed into T scores, and the T scores equal to or above 63 will be considered indicative of clinically significant symptomatology.
Change in the intestinal permeabily parameters of sugar absorption test | Before the start of the study (time 0) and after 90 days of treatment (time 90).
  For the evaluation of intestinal permeability, a test solution is prepared with 40 g sucrose (Su), 10 g lactulose (La) and 5 g mannitol (Ma) dissolved in 100 ml of water.
  The participants drink the test solution in the morning after an overnight fast, and all urine samples are collected for the subsequent 5 h. Urine samples were stored at -80°C until analysis. The detection and measurement of the three sugar probes, Su, La, and Ma in urine are performed by high-performance anion-exchange chromatography coupled with pulsed amperometric detection. Su, La, and Ma will be expressed as the percentage of excretion of the ingested amount of sugars. La and Ma measurements will then be reported as a ratio (La/Ma) to evaluate the permeability of the small intestinal tract.
Change in the markers of integrity of the intestinal barrier | Before the start of the study (time 0) and after 90 days of treatment (time 90).
  To evaluate intestinal barrier markers, blood samples are collected in ice chilled tubes containing Aprotinin and EDTA. The separated plasma are stored at -70 °C until assay. Serum levels of zonulin, IFABp, DAO, copeptin, meteorin, somatostatin and serotonin, are measured by enzyme immunoassay technique using commercial kits before and after the dietary interventions. All these parameters provide information about the state of health of the intestinal mucosa and will be expressed as ng/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Russo, MD, Principal Investigator — National Institute for Digestive Diseases IRCCS " Saverio de Bellis"
Locations (1):
- IRCCS Saverio de Bellis, Castellana Grotte, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tuck CJ, Reed DE, Muir JG, Vanner SJ. Implementation of the low FODMAP diet in functional gastrointestinal symptoms: A real-world experience. Neurogastroenterol Motil. 2020 Jan;32(1):e13730. doi: 10.1111/nmo.13730. Epub 2019 Sep 30. PMID 31571351
- [Background] Linsalata M, Riezzo G, Orlando A, D'Attoma B, Prospero L, Tutino V, Notarnicola M, Russo F. The Relationship between Low Serum Vitamin D Levels and Altered Intestinal Barrier Function in Patients with IBS Diarrhoea Undergoing a Long-Term Low-FODMAP Diet: Novel Observations from a Clinical Trial. Nutrients. 2021 Mar 21;13(3):1011. doi: 10.3390/nu13031011. PMID 33801020
- [Background] Orlando A, Tutino V, Notarnicola M, Riezzo G, Linsalata M, Clemente C, Prospero L, Martulli M, D'Attoma B, De Nunzio V, Russo F. Improved Symptom Profiles and Minimal Inflammation in IBS-D Patients Undergoing a Long-Term Low-FODMAP Diet: A Lipidomic Perspective. Nutrients. 2020 Jun 2;12(6):1652. doi: 10.3390/nu12061652. PMID 32498383
- [Background] Avila CM, Rodriguez-Suarez C, Atienza SG. Tritordeum: Creating a New Crop Species-The Successful Use of Plant Genetic Resources. Plants (Basel). 2021 May 20;10(5):1029. doi: 10.3390/plants10051029. PMID 34065483
- [Background] Vaquero L, Comino I, Vivas S, Rodriguez-Martin L, Gimenez MJ, Pastor J, Sousa C, Barro F. Tritordeum: a novel cereal for food processing with good acceptability and significant reduction in gluten immunogenic peptides in comparison with wheat. J Sci Food Agric. 2018 Apr;98(6):2201-2209. doi: 10.1002/jsfa.8705. Epub 2017 Nov 9. PMID 28963718
- [Background] Rotondi Aufiero V, Fasano A, Mazzarella G. Non-Celiac Gluten Sensitivity: How Its Gut Immune Activation and Potential Dietary Management Differ from Celiac Disease. Mol Nutr Food Res. 2018 May;62(9):e1700854. doi: 10.1002/mnfr.201700854. Epub 2018 Apr 20. PMID 29578652
- [Background] Barmeyer C, Schumann M, Meyer T, Zielinski C, Zuberbier T, Siegmund B, Schulzke JD, Daum S, Ullrich R. Long-term response to gluten-free diet as evidence for non-celiac wheat sensitivity in one third of patients with diarrhea-dominant and mixed-type irritable bowel syndrome. Int J Colorectal Dis. 2017 Jan;32(1):29-39. doi: 10.1007/s00384-016-2663-x. Epub 2016 Sep 30. PMID 27695975
- [Background] Russo F, Riezzo G, Linsalata M, Orlando A, Tutino V, Prospero L, D'Attoma B, Giannelli G. Managing Symptom Profile of IBS-D Patients With Tritordeum-Based Foods: Results From a Pilot Study. Front Nutr. 2022 Feb 15;9:797192. doi: 10.3389/fnut.2022.797192. eCollection 2022. PMID 35242794